CLINICAL TRIAL: NCT03156413
Title: The Evaluation of a Nasal Mask for the Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-206
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Sleep Disordered Breathing; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- F&P Nasal Mask (Experimental): Trial nasal pillows CPAP mask
  Interventions: Device: F&P nasal mask

INTERVENTIONS:
Device: F&P nasal mask — Investigative Nasal Mask to be used for OSA therapy

SUMMARY:
This investigation is designed to evaluate the performance as well as the patients overall acceptance of the mask.

DETAILED DESCRIPTION:
A maximum of 12 OSA participants who currently use a nasal mask will be recruited for the trial. Participant will be on the trial for 1 night (in-lab)

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years of age)
* Able to give consent
* Apnea hypopnea Index (AHI)≥ 5 on diagnostic night
* Prescribed PAP for OSA
* Existing nasal mask user

Exclusion Criteria:

* Inability to give consent
* Patients who are in a coma or a decreased level of consciousness
* Anatomical or physiological conditions making automatic positive airway pressure (APAP) therapy inappropriate (e.g. unconsolidated facial structure)
* Commercial drivers who are investigated by New Zealand Transport Agency
* Current diagnosis of carbon dioxide (CO2) retention
* Pregnant or may think they are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-06-05 (Actual)

PRIMARY OUTCOMES:
Ease of use | 1 night
  Subjective questionnaire
Acceptability | 1 night
  Subjective questionnaire

SECONDARY OUTCOMES:
Objective leak data | 1 night
  Data obtained from participant's device - Objective

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Gunson, Principal Investigator — Sponsor Employee
Locations (1):
- Fisher and Paykel Healthcare, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No
For product development purposes only. Data will be deidentified.